CLINICAL TRIAL: NCT03905824
Title: Randomized, Multicentric, Prospective, Double-blind Study: Effectiveness of Adding Allogenic Stem Cells to a Platelet-poor Plasma Scaffold After Arthroscopic Debridement and Microfractures in Patients With Osteochondral Lesions of the Talus
Brief Title: The Effectiveness of Adding Allogenic Stem Cells After Traditional Treatment of Osteochondral Lesions of the Talus
Acronym: OLT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Manuel J Pellegrini, Principal Investigator, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OLT Protocol
Record Dates: First submitted 2019-03-29; First posted 2019-04-05 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Osteochondral Fracture of Talus
MeSH Terms: interventions — Debridement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Debridement and microfracture in LOC + Cells (Experimental): Traditional debridement and microfracture treatment adding a platelet-poor plasma (PPP) scaffold embedded in allogenic stromal mesenchymal cells derived from the umbilical cord in patients with osteochondral lesions of the talus.
  Interventions: Biological: Allogenic stromal mesenchymal cells derived from the umbilical cord; Procedure: Debridement and microfracture
- Debridement and microfracture in LOC (Active Comparator): Traditional debridement and microfracture treatment in patients with osteochondral lesions of the talus.
  Interventions: Procedure: Debridement and microfracture

INTERVENTIONS:
Biological: Allogenic stromal mesenchymal cells derived from the umbilical cord — Platelet-poor plasma (PPP) scaffold embedded in allogenic stromal mesenchymal cells derived from the umbilical cord added to the traditional treatment for osteochondral lesions of the talus
  Arms: Debridement and microfracture in LOC + Cells
Procedure: Debridement and microfracture — Debridement and microfracture in LOC is the traditional treatment for osteochondral lesions of the talus

SUMMARY:
Randomized, multicentric, prospective, double-blind study: effectiveness of adding allogenic stem cells to a platelet-poor plasma scaffold after arthroscopic debridement and microfractures in patients with osteochondral lesions of the talus Osteochondral lesions of the talus (LOC), affects the ankle cartilage, which it seems to have less repair capacity than that of other joints such as the knee of the hip. The LOC can be an important source of pain and affects comparatively younger, working age and athletically active patients.

Although there are several therapeutic strategies, debridement and microfractures performed arthroscopically are the most frequent procedures. After this surgery, it is expected that fibrocartilage will form that covers the osteochondral lesion. Though good results have been reported, this fibrocartilage presents histological characteristics of lower quality to those of the native articular cartilage.

Based on previous studies in different joints, it is hypothesized that the augmentation treatment of osteochondral lesions of the talus with mesenchymal allogeneic stromal cells derived from the umbilical cord produces better clinical and imaging results than standard treatment with debridement and microfractures only.

Therefore, the present study seeks to compare the effectiveness of traditional debridement and microfracture treatment versus adding a platelet-poor plasma (PPP) scaffold embedded in allogeneic mesenchymal stromal cells derived from the umbilical cord in patients with osteochondral lesions of the talus.

DETAILED DESCRIPTION:
As with other major joints of the lower limb that carry weight (hip, knee), the osteochondral lesion (LOC) of the talus, can be a major source of pain and disability for the affected patient. The LOC of the talus can appear after one (or repeated) traumatic injury, compromises the bone and adjacent cartilage, being able to cause blisters in the cartilage layers, lesions similar to a cyst within the bone under the cartilage, or fracture of the cartilage and the bony layers.

The ankle joint supports multiple loads of the corporal weight in the daily activities, the reason why the properties of the cartilage in the ankle are different from those that appear in the hip and the knee. In the absence of an injury, the cartilage of the ankle has better resistance and tension properties to face the increase of forces than the hip or knee throughout life.

However, once an injury appears, the cartilage of the ankle appears to have less repair capacity compared to the hip or knee. Since the most common cause of LOC of the talus is post-traumatic, the average age of these patients is comparatively lower than that of patients affected by injuries to other joints.

Osteochondral injuries have an incidence of 27 per 10,0000 inhabitants in the USA. They are injuries that usually affect the working population and active sportsperson, producing pain, functional limitation and that probably contribute towards the evolution of an accelerated joint degeneration. Currently, there are multiple treatment modalities used by ankle and foot surgeons. These include debridement and microfractures of the subchondral plaque, utilization of totipotential cells, osteochondral autograft/allograft, tibiotalar arthrodesis, and partial/total ankle arthroplasty. However, no treatment offers a clear superiority over the others.

Debridement and microfractures performed arthroscopically is the most frequently used procedure and involves; the removal of degenerated cartilage and subchondral bone; obtaining firm lesional edges that prevent the spread of the lesion; and finally the stimulation of the bone marrow talar by performing microfractures of the subchondral plate. This with the hope that fibrocartilage will form that covers the osteochondral lesion. Although this fibrocartilage has histological characteristics different from those of native articular cartilage, good results have been reported in 82% of the cases when combining good quality studies in this regard.

The standard technique is not able to generate a replacement articular cartilage strong enough to support the joint loads to which the ankle is exposed. Therefore, clinical trials seek to increase the traditional treatment of debridement and microfractures with the intra-articular use of totipotent cells at the end of the procedure. Although the results of these series are promising and comparable at least to those of traditional treatment, the absence of comparative studies between them complicates the choice of treatment for both the patient and the surgeon. For this reason, the investigators have designed a prospective, comparative, double-blind study that will allow elucidating which of these interventions is the best alternative for our patients.

General Objective:

To compare the effectiveness of traditional debridement and microfracture treatment versus adding a platelet-poor plasma (PPP) scaffold embedded in allogenic stromal mesenchymal cells derived from the umbilical cord in patients with osteochondral lesions of the talus.

Specific Objectives:

* To compare functional and radiological results before versus post-surgery within each group studied (control and experimental)
* To compare functional results after surgery of the groups in traditional treatment versus traditional treatment plus mesenchymal stromal cells (MSC).
* To compare the quality of repair of the tissues of the groups in traditional treatment versus traditional treatment plus mesenchymal stromal cells (MSC).

Work hypothesis:

The augmentation treatment of the osteochondral lesions of the talus with mesenchymal cells produces better clinical and imaging results than standard treatment with only debridement and microfractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a symptomatic osteochondral lesion of the Talus.
* Magnetic resonance of the ankle showing osteochondral injury of a single talus, with perilesional oedema

Exclusion Criteria:

* Recurrent osteochondral lesions of the talus
* Multiple osteochondral lesions
* Severe ankle instability, requiring open repair
* History of a previous foot or ankle surgery of the ipsilateral foot
* Rheumatoid arthritis
* Inability to return to the surgery site to practice long-term follow-up evaluations or lack of readiness to complete the indicated evaluation forms.
* Patients with a qualitative or quantitative commitment that prevents consent or assent their participation in the study.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change on tissue reparation quality | Baseline and 1 year follow up
  Magnetic resonance observation of cartilage repair tissue (MOCART). The MOCART classification is one of the most frequently used MR score for postoperative cartilage repair tissue evaluation. The MOCART score is a 9-part and 29-item scoring system, also resulting in a final cartilage repair tissue score between 0 and 100 points; 0 points represent the worst imaginable score, 100 points represent the best imaginable score.
Change over time of general health status | Baseline, 1 year and 2 years follow up
  The MOS SF-36, It is a generic scale to evaluate health/disease status. It comprises 36 items divided into two components: Physical Health (PH) and Mental Health (MH). PH includes four subscales: Physical Function (PF), Role Physical (RP), Bodily Pain (BP), and General Health (GH). MH includes four subscales: Vitality (V), Social functioning (SF), Role Emotional (RE), and General Health (GH).
  Each component (PH and MH) and each of the eight subscale scores are transformed into a 0-to-100 scale. Higher scores represent better health status
Change over time of functional limitations of foot and ankle. | Baseline, 1 year and 2 years follow up
  The Foot and Ankle Outcome Score (FAOS) evaluates functional limitations related to foot and ankle issues. Consist in 42 items that cover 5 dimensions: Symptoms (S: 7 items), Pain (P: 9 items), Activities of Daily Living (ADL: 17 items), Sport and Recreation Activities (SRA: 5 items), and foot and ankle related Quality of Life (QoL: 4 items). Raw scores of each sub-scales results of the sum of each item score.
  These raw scores are standardised into a 0 to 100 scale; higher scores mean higher dysfunction due to foot/ankle condition.
Change over time of functionality of musculoskeletal ankle and foot pathology | Baseline, 1 year and 2 years follow up
  The Foot and Ankle Ability Measure (FAAM) scale aims to evaluate overtime changes in the functionality of the same patient in musculoskeletal ankle and foot pathology. It is a survey that consists of 21 items about activities of daily living, and 8 items about sports skills.
  Raw scores of each sub-scales are standardised into a 0 to 100 scale; higher scores mean higher dysfunction due to foot/ankle condition.
Change on declared pain | Baseline, 1 year and 2 years follow up
  Visual Analog Scale for Pain (VAS-Pain): a pain rating scale based on self-reported measures of symptoms. A 10cm line numbered from 0 to 10 represents a continuum between "no pain" (zero) and "worst pain" (ten).
  It can also be interpreted as a 0-to-100 points score.

SECONDARY OUTCOMES:
Surgical time | During surgery
  Duration (in minutes) of the surgery
Complication rate | Two years follow up from baseline (surgery)
  Including the number of participants with:
  * post-surgery infections
  * temporal or permanent damage of nerve as a result of pressure or hematoma
  * with venose thrombosis, pulmonary embolism or heart stroke
Cost-effective comparative analysis | Two years follow up from baseline (surgery)
  Comparison of the overall costs and results of both groups

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Pellegrini, MD, Principal Investigator — Universidad de Chile Clinical Hospital
Locations (1):
- Universidad de Chile Clinical Hospital, Santiago, Independencia, Chile

IPD SHARING:
Plan to Share IPD: No